CLINICAL TRIAL: NCT05411731
Title: Effect of Modified Constraint Induced Movement Therapy on Range of Motion, Function and Disability in Children With Obstetric Brachial Plexus Injury
Brief Title: Modified Constraint Induced Movement Therapy in Children With Obstetric Brachial Plexus Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/22/0701
Record Dates: First submitted 2022-06-06; First posted 2022-06-09 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Obstetric; Injury
Keywords: birth injuries therapy; arm function; constraint induced movement therapy; brachial plexus neuropathies
MeSH Terms: conditions — Wounds and Injuries; Brachial Plexus Neuropathies | interventions — Constraint Induced Movement Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional physical therapy treatment (Active Comparator): Patients in this group will receive conventional physical therapy i.e. stretching, strengthening exercises, Aeroplan positioning
  Interventions: Other: Conventional physical therapy treatment
- Constraint induced movement therapy (Experimental): patients of this group will receive the same treatment along with constraint induced movement therapy
  Interventions: Other: Constraint induced movement therapy

INTERVENTIONS:
Other: Conventional physical therapy treatment — The control group (group A) will receive the exercise program which focused on improving the arm function as well as shoulder abduction and external rotation for 10 week.
  stretching Aeroplan positioning
  Arms: Conventional physical therapy treatment
Other: Constraint induced movement therapy — The study group (group B) who will receive Modified constraint induced movement therapy for 3 hrs. a day 12 hrs. a week in addition to the same exercise program given to the control group for 10 weeks.
  Arms: Constraint induced movement therapy

SUMMARY:
The aim of this study was to increase and improve the use of affected extremity in obstetric brachial plexus palsy children while restricting the use of less affected arm and the purpose was to improve the function, Range of motion and disability in affected arm of children with brachial plexus injury.

ELIGIBILITY:
Inclusion Criteria:

* 3 to 10 years
* Both genders will be included
* Deficiency of shoulder abduction and external rotation
* Who can follows command

Exclusion Criteria:

* uncontrolled seizures
* Orthopedic and/or neurological surgery.
* A visual impairment interfering with treatment/testing.
* Unable to actively engage in assessment process

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2022-04-30 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Mallet grading system | 4 weeks
  The Mallet grading system is a commonly used functional scoring system to assess shoulder abduction/external rotation deficits in children with obstetric brachial plexus palsy. One feature of the Mallet score is that each grade is translated in to certain degree of deficiencies in both shoulder abduction and external rotation. A scale of 1 to 5 is used to evaluate shoulder abduction, global external rotation, and hand to neck, hand to back, and hand to mouth positions.

SECONDARY OUTCOMES:
goniometer | 4th week
  changes from the baseline ROM of shoulder abduction and external rotation as well as elbow ranges was measured by goniometer was measured by can evaluate both active as well as passive range of motion.
Upper extremity function index | 4th week
  It is a self-administered questionnaire which measures disability in people with upper extremity orthopaedic conditions. The questionnaire lists 20 activities and the patient gives a score to each based on the difficulty they have completing that activity. It is evaluated on a 5-point scale that refers to the perceived difficulty in performing the mentioned action:
  * Extreme difficulty or unable to perform activity (0 points);
  * Quite a bit of difficulty (1 point);
  * Moderate difficulty (2 points);
  * A little bit of difficulty (3 points);
  * No difficulty (4 points).
  The overall Upper extremity function index (UEFI) result ranges between 0 and 80, where 0 indicates most severe limitation and 80 suggests least limitation. Changes from baseline function of affected extremity was given by this tool.

CONTACTS AND LOCATIONS:
Overall Officials: Hafiza Mehjabeen, ppdpt, Principal Investigator — Riphah International University
Locations (1):
- Bakhtawar Amin Trust Teaching Hospital, Multan Khurd, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pejkova S, Filipce V, Peev I, Nikolovska B, Jovanoski T, Georgieva G, Srbov B. Brachial Plexus Injuries - Review of the Anatomy and the Treatment Options. Pril (Makedon Akad Nauk Umet Odd Med Nauki). 2021 Apr 23;42(1):91-103. doi: 10.2478/prilozi-2021-0008. PMID 33894122
- [Background] Souza L, Lustosa L, Silva AEL, Martins JV, Pozzo T, Vargas CD. Kinematic Changes in the Uninjured Limb After a Traumatic Brachial Plexus Injury. Front Hum Neurosci. 2021 Dec 9;15:777776. doi: 10.3389/fnhum.2021.777776. eCollection 2021. PMID 34955793
- [Background] Adler JB, Patterson RL Jr. Erb's palsy. Long-term results of treatment in eighty-eight cases. J Bone Joint Surg Am. 1967 Sep;49(6):1052-64. No abstract available. PMID 6038856
- [Background] Sparrow J, Zhu L, Gajjar A, Mandrell BN, Ness KK. Constraint-Induced Movement Therapy for Children With Brain Tumors. Pediatr Phys Ther. 2017 Jan;29(1):55-61. doi: 10.1097/PEP.0000000000000331. PMID 27984470
- [Background] Eren B, Karadag Saygi E, Tokgoz D, Akdeniz Leblebicier M. Modified constraint-induced movement therapy during hospitalization in children with perinatal brachial plexus palsy: A randomized controlled trial. J Hand Ther. 2020 Jul-Sep;33(3):418-425. doi: 10.1016/j.jht.2019.12.008. Epub 2020 Mar 7. PMID 32151503
- [Background] Berggren J, Baker LL. Therapeutic application of electrical stimulation and constraint induced movement therapy in perinatal brachial plexus injury: A case report. J Hand Ther. 2015 Apr-Jun;28(2):217-20; quiz 221. doi: 10.1016/j.jht.2014.12.006. Epub 2014 Dec 17. PMID 25841560
- [Background] Wang Q, Zhao JL, Zhu QX, Li J, Meng PP. Comparison of conventional therapy, intensive therapy and modified constraint-induced movement therapy to improve upper extremity function after stroke. J Rehabil Med. 2011 Jun;43(7):619-25. doi: 10.2340/16501977-0819. PMID 21603848
- [Background] El-Shamy S, Alsharif R. Effect of virtual reality versus conventional physiotherapy on upper extremity function in children with obstetric brachial plexus injury. J Musculoskelet Neuronal Interact. 2017 Dec 1;17(4):319-326. PMID 29199193
- [Background] Zielinski IM, van Delft R, Voorman JM, Geurts ACH, Steenbergen B, Aarts PBM. The effects of modified constraint-induced movement therapy combined with intensive bimanual training in children with brachial plexus birth injury: a retrospective data base study. Disabil Rehabil. 2021 Aug;43(16):2275-2284. doi: 10.1080/09638288.2019.1697381. Epub 2019 Dec 8. PMID 31814455
- [Background] Ramey SL, DeLuca SC, Stevenson RD, Conaway M, Darragh AR, Lo W; CHAMP. Constraint-Induced Movement Therapy for Cerebral Palsy: A Randomized Trial. Pediatrics. 2021 Nov;148(5):e2020033878. doi: 10.1542/peds.2020-033878. Epub 2021 Oct 14. PMID 34649982
- [Background] Werner JM, Berggren J, Loiselle J, Lee GK. Constraint-induced movement therapy for children with neonatal brachial plexus palsy: a randomized crossover trial. Dev Med Child Neurol. 2021 May;63(5):545-551. doi: 10.1111/dmcn.14741. Epub 2020 Nov 21. PMID 33219706